CLINICAL TRIAL: NCT01414205
Title: An Open-label, Multicenter, Randomized Phase II Trial Comparing the Efficacy, Safety, and Pharmacokinetics of GA101 1000 mg Versus 2000 mg in Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study Comparing Obinutuzumab (RO5072759; GA101) 1000 Milligram (mg) Versus 2000 mg in Participants With Previously Untreated Chronic Lymphocytic Leukemia (CLL) (GAGE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAO4768g; GO25677 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; Adrenal Cortex Hormones

ARMS (2):
- Obinutuzumab 1000 mg (Experimental): Participants received a 1000 mg intravenous (IV) infusion, on days 1 (split dose 100 mg on Day 1 and 900 mg on Day 2), 8 and 15 of cycle 1 and day 1 of cycles 2 - 8, 21 day cycles. All participants received corticosteroids IV prior to the initial dose.
  Interventions: Drug: Obinutuzumab; Drug: Corticosteroids
- Obinutuzumab 2000 mg (Experimental): Participants received a 2000 mg IV infusion, on days 1 (split dose 100 mg Day 1, 900 mg Day 2 and 1000 mg Day 3), 8 and 15 of cycle 1 and day 1 of cycles 2 -8, 21 day cycles. All participants received corticosteroids IV prior to the initial dose.
  Interventions: Drug: Obinutuzumab; Drug: Corticosteroids

INTERVENTIONS:
Drug: Obinutuzumab — Participants were administered obinutuzumab either at 1000 mg or 2000 mg on Day 1, 8, 15 of Cycle 1 and then on Day 1 of each 21 day cycles for up to 8 cycles.
  Other Names: RO5072759; GA101
Drug: Corticosteroids — Participants were administered corticosteroids IV prior to the initial dose.

SUMMARY:
This open-label, multicenter, randomized study compared the efficacy, safety and pharmacokinetics of obinutuzumab (RO5072759; GA101) 1000 mg versus 2000 mg in participants with previously untreated CLL. Participants were randomized to receive a maximum of 8 cycles (28-day cycle) of obinutuzumab (1000 mg intravenous [IV] infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of each subsequent cycle up to 8 cycles or maximum of 8 cycles of obinutuzumab (2000 mg IV infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of each subsequent cycle up to 8 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CD20-positive B-cell CLL (per International Workshop on Chronic Lymphocytic Leukemia [IWCLL] guidelines)
* Rai Stage III/IV or Binet Stage C disease, or Rai Stage I/II or Binet Stage B disease that requires treatment according to IWCLL guidelines
* No previous treatment for CLL chemotherapy, radiotherapy or immunotherapy; no previous rituximab treatment for autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP); prior use of steroids for AIHA or ITP is allowed
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2

Exclusion Criteria:

* Confirmed diagnosis of Transformation of CLL to aggressive B-cell malignancy
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Evidence of severe, uncontrolled concomitant disease
* Known active infection or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks before the start of Cycle 1
* Seropositive for human immunodeficiency virus (HIV)
* Positive for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology)
* Positive for hepatitis C (hepatitis C virus [HCV] antibody serology testing)
* Pregnant or lactating women
* Concurrent (or within 7 days prior to first dose of study treatment) systemic corticosteroid use, except for low-dose corticosteroid therapy used to treat chronic medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (31):
  - Univ of Alabama at Birmingham; UAB Comprehensive Cancer Ctr, Birmingham, Alabama
  - Arizona Oncology, Tucson, Arizona
  - Arizona Clinical Research Ctr, Tucson, Arizona
  - University of California; Moores Cancer Center, La Jolla, California
  - USC Norris Cancer Center, Los Angeles, California
  - USC/Norris Can Ctr; IDS Pharm, Los Angeles, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical Group, Pasadena, California
  - Univ of Colorado Canc Ctr, Aurora, Colorado
  - Rocky Mountain Cancer Center; Medical Oncology, Denver, Colorado
  - Kootenai Cancer Center, Post Falls, Idaho
  - Goshen Hlth Sys Ctr Can Care, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Purchase Cancer Group, Paducah, Kentucky
  - Hem Onc Assoc of Northern NJ; Carol G. Simon Canc Ctr, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Mark H. Zangmeister Center, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - INTEGRIS Cancer Inst of OK, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Ctr - 520 Country Club, Eugene, Oregon
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - US Oncology Research Pharm., Fort Worth, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - SW Virginia Hem Onc, Roanoke, Virginia
  - Shenandoah Oncology Associates, Winchester, Virginia
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- [Derived] Byrd JC, Flynn JM, Kipps TJ, Boxer M, Kolibaba KS, Carlile DJ, Fingerle-Rowson G, Tyson N, Hirata J, Sharman JP. Randomized phase 2 study of obinutuzumab monotherapy in symptomatic, previously untreated chronic lymphocytic leukemia. Blood. 2016 Jan 7;127(1):79-86. doi: 10.1182/blood-2015-03-634394. Epub 2015 Oct 15. PMID 26472752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Started | 41 | 39
Received Study Drug | 40 | 38
Completed | 34 | 32
Not Completed | 7 | 7
Not completed — Death | 5 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Randomized but not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (10.0) | 64.3 (12.4) | 65.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with complete response (CR), CR with incomplete marrow recovery (CRi) or partial response (PR) as assessed by the investigator according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) guidelines two months after last treatment. CR required: blood lymphocytes < 4 x 10^9/Liter (L), absence of lymphadenopathy (≤ 1.5 centimeter (cm) in long axis by Computed Tomography), no hepatomegaly or splenomegaly, absence of disease, Neutrophils > 1.5 x 10^9/L, Platelets > 100 x 10^9/L, Hemoglobin >11 g/dL, bone marrow normal and lymphoid nodules absent. CRi was CR with incomplete marrow recovery. PR required: 50% decrease in peripheral blood lymphocyte count, 50% reduction in lymphadenopathy, 50% reduction of liver and/or spleen enlargement if enlarged at baseline, Neutrophils > 1.5 x 10^9/L or > 50% of pretreatment value, Platelets > 100 x 10^9/L or 50% of pretreatment value and Hemoglobin > 11 g/dL or > 50% of pretreatment value.
Time Frame: Week 32
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 41 | 39
Percentage of participants | 48.8 | 66.7
Statistical Analysis 1: Comparison: Obinutuzumab 1000 mg vs Obinutuzumab 2000 mg; Test type: Superiority or Other; p = 0.0779, Cochran-Mantel-Haenszel; P-values based on stratified Cochran-Mantel-Haenszel test by the randomization stratification factors as supportive analyses; Difference (Hauck-Anderson) = 17.89, 95% CI 2-sided [-4.95 to 40.72]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the randomization to the first occurrence of progression or death, whichever occurred first.
Time Frame: Up to 4 years, 5 months
Population: Intent-to-treat population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 41 | 39
Months | 25.2 [15.9 to 30.4] | 26.0 [20.2 to 34.2]

3. Secondary Outcome: Duration of Response
Time Frame: Up to 4 years, 5 months
Population: Duration of response was not analyzed as investigators did not perform response assessments at regular intervals during the follow-up period.
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants Surviving at End-of-Study
Time Frame: Up to 4 years, 5 months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Participants
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 41 | 39
Participants | 35 | 37

5. Secondary Outcome: Percentage of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution. A SAE was any AE that was one of the following: fatal, life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product or considered a significant medical event by the investigator. Additional information about AEs can be found in the Adverse Event Section.
Time Frame: Up to 4 years, 5 months
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 40 | 38
Percentage of participants
  Adverse Events | 100.0 | 100.0
  Serious Adverse Events | 20.0 | 21.1

6. Secondary Outcome: Percentage of Participants With Adverse Events of Interest
Description: Adverse Events of interest for this study were: serious infusion related reactions during or within 24 hours of infusion, serious neutropenia, serious infection, tumor lysis syndrome and Hepatitis B reactivation.
Time Frame: Up to 4 years, 5 months
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 40 | 38
Percentage of participants
  Serious Infusion-Related Reactions (IRR) | 7.5 | 5.3
  Serious Neutropenia | 5.0 | 5.3
  Serious Infection | 5.0 | 5.3
  Tumor Lysis Syndrome | 0.0 | 2.6
  Hepatitis B Reactivation | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Study Discontinuation
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution.
Time Frame: Up to 4 years, 5 months
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 40 | 38
Percentage of participants | 0 | 0

8. Secondary Outcome: PK Parameter: Maximum Serum Concentration (Cmax)
Description: Blood was collected for Pharmacokinetic (PK) Parameter Cmax after dose administration on Day 1 of Cycle 8. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA) measured in micrograms per milliliter (μg/mL).
Time Frame: Day 148 (at end of infusion)
Population: All randomized participants who received study drug with PK data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 37 | 33
μg/mL | 600 (45.6) | 1190 (34.9)

9. Secondary Outcome: PK Parameter: Area Under the Serum Concentration-Time Curve Between Dosing Interval Tau (AUCt )
Description: Blood was collected for PK Parameters before and after dose administration on Day 1 of Cycle 8. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA) measured in day times micrograms per milliliter (day*μg/mL).
Time Frame: Day 148 (pre-infusion, at end of infusion, 5, 8 and 12 days after start of infusion)
Population: All randomized participants who received study drug with PK data available for analysis. Participants with insufficient data points for PK estimation were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 26 | 25
day*μg/mL | 8230 (58.3) | 16500 (50.3)

10. Secondary Outcome: PK Parameter: Clearance at Steady State (CLss)
Description: Blood was collected for PK Parameters before and after dose administration on Day 1 of Cycle 8. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). CLss is reported in milliliters per day (mL/day).
Time Frame: Day 148 (pre-infusion, at end of infusion, 5, 8 and 12 days after start of infusion)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 26 | 25
mL/day | 121 (58.3) | 122 (50.3)

11. Secondary Outcome: PK Parameter: Volume of Distribution at Steady State (Vss)
Description: Blood was collected for PK Parameters before and after dose administration on Day 1 of Cycle 8. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). Vss is reported in liters.
Time Frame: Day 148 (pre-infusion, at end of infusion, 5, 8 and 12 days after start of infusion)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 24 | 23
Liters | 7.08 (73.2) | 6.68 (74.7)

12. Secondary Outcome: PK Parameter: Terminal Half-Life (t1/2)
Description: Blood was collected for PK Parameters before and after dose administration on Day 1 of Cycle 8. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). T1/2 was reported in Days.
Time Frame: Day 148 (pre-infusion, at end of infusion, 5, 8 and 12 days after start of infusion)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 24 | 23
Days | 30.6 (87.1) | 26.3 (80.1)

13. Secondary Outcome: PK: Serum Concentrations of Obinutuzumab (Follow-Up Visits)
Description: Blood serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA) measured in micrograms per milliliter (μg/mL).
Time Frame: Months 3, 6, 9, and 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 37 | 33
μg/mL
  Month 3 (n=14, 10) | 41.2 (63.3) | 98.9 (88.9)
  Month 6 (n=19, 15) | 15 (21.4) | 12.6 (17.7)
  Month 9 (n=24, 23) | 2.63 (4.4) | 4.09 (9.42)
  Month 12 (n=16, 18) | 0.633 (1.11) | 0.857 (1.74)

14. Secondary Outcome: Pharmacodynamics: Number of Participants With Peripheral Blood B-cell Depletion
Description: Blood was sent to a central laboratory for the evaluation of cluster of differentiation 19 (CD19) by flow cytometry. B-cell depletion was defined as a CD19 result < 0.07 × 10^9/L after at least one dose of study drug has been administered.
Time Frame: Up to 4 years, 5 months
Population: Participants from the Safety Evaluable Population, all randomized participants who received at least one dose of study drug, who had data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 40 | 38
Participants
  At Last Antibody Administration (n=40, 38) | 31 | 31
  Up to 6 Months of Follow-Up (FU) (n=30, 31) | 28 | 28
  Within 6-12 Months of Follow-up (n=24, 24) | 16 | 17
  Within 12-18 Months of Follow-up (n=17, 17) | 11 | 9
  Within 18-24 Months of Follow-up (n=10, 9) | 5 | 8
  Within 24-30 Months of Follow-up (n=4, 6) | 2 | 5
  Within 30-36 Months of Follow-up (n=1, 3) | 1 | 3
  Within 36-42 Months of Follow-up (n=0, 0) | 0 | 0
  After 42 Months of Follow-up (n=0, 0) | 0 | 0

15. Secondary Outcome: Pharmacodynamics: Number of Participants With Peripheral Blood B-cell Recovery
Description: Blood was sent to a central laboratory for the evaluation of cluster of differentiation 19 (CD19) by flow cytometry. B-cell recovery was defined as a CD19 result ≥ 0.07 × 10^9/L, where CD19 was previously depleted. B-cell recovery was only considered possible following the last dose of study treatment. The number of participants with B-cell recovery from End of Treatment to 6 months of Follow-up is reported in two categories: Recovery with Progressive Disease (PD) [PD before B-cell recovery or PD within 45 days after recovery] or Recovery without PD. PD required one of the following: 50% increase in the absolute number of circulating lymphocytes, Appearance of new palpable lymph nodes, 50% increase in the longest diameter of any previous site of lymphadenopathy, 50% increase in the enlargement of the liver and/or spleen or Transformation to a more aggressive histology.
Time Frame: Up to 4 years, 5 months
Population: Participants from the Safety Evaluable Population, all randomized participants who received at least one dose of study drug, with B-Cell depletion.
Measure: Number; unit: Participants
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Number analyzed (Participants) | 40 | 38
Participants
  Up to 6 Months FU: Recovery with PD (n=30, 31) | 0 | 0
  Up to 6 Months FU: Recovery without PD (n=30, 31) | 2 | 3
  6-12 Months FU: Recovery with PD (n=24, 24) | 1 | 0
  6-12 Months FU: Recovery without PD (n=24, 24) | 7 | 7
  12-18 Months FU: Recovery with PD (n=17, 17) | 0 | 0
  12-18 Months FU: Recovery without PD (n=17, 17) | 6 | 8
  18-24 Months FU: Recovery with PD (n=10, 9) | 0 | 0
  18-24 Months FU: Recovery without PD (n=10, 9) | 5 | 1
  24-30 Months FU: Recovery with PD (n=4, 6) | 0 | 0
  24-30 Months FU: Recovery without PD (n=4, 6) | 2 | 1
  30-36 Months FU: Recovery with PD (n=1, 3) | 0 | 0
  30-36 Months FU: Recovery without PD (n=1, 3) | 0 | 0
  36-42 Months FU: Recovery with PD (n=0, 0) | 0 | 0
  36-42 Months FU: Recovery without PD (n=0, 0) | 0 | 0
  After 42 Months FU: Recovery with PD (n=0, 0) | 0 | 0
  After 42 Months FU: Recovery without PD (n=0, 0) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 years, 5 months
Arm/Group | Obinutuzumab 1000 mg | Obinutuzumab 2000 mg
Serious Adverse Events (participants affected / at risk) | 8/40 | 8/38
Other Adverse Events (participants affected / at risk) | 40/40 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab 1000 mg (N=40) | Obinutuzumab 2000 mg (N=38)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab 1000 mg (N=40) | Obinutuzumab 2000 mg (N=38)
Infusion related reaction (Injury, poisoning and procedural complications) | 30 | 24
Pyrexia (General disorders) | 16 | 18
Fatigue (General disorders) | 16 | 12
Chills (General disorders) | 8 | 7
Oedema peripheral (General disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 15 | 10
Vomiting (Gastrointestinal disorders) | 11 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Constipation (Gastrointestinal disorders) | 3 | 5
Dizziness (Nervous system disorders) | 10 | 7
Headache (Nervous system disorders) | 11 | 4
Neutropenia (Blood and lymphatic system disorders) | 14 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 7
Anaemia (Blood and lymphatic system disorders) | 7 | 3
Flushing (Vascular disorders) | 8 | 9
Hypotension (Vascular disorders) | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 6 | 7
Chest discomfort (General disorders) | 3 | 4
Asthenia (General disorders) | 3 | 0
Influenza like illness (General disorders) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Laceration (Injury, poisoning and procedural complications) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 2 | 3
Tremor (Nervous system disorders) | 2 | 2
Memory impairment (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 2 | 2
Fungal skin infection (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 2 | 0
Depression (Psychiatric disorders) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 1 | 2
Visual impairment (Eye disorders) | 1 | 2
Nocturia (Renal and urinary disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Blood magnesium decreased (Investigations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2
Chest Pain (General disorders) | 2 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vision Blurred (Eye disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.